CLINICAL TRIAL: NCT02714192
Title: Evaluation of the Safety of Exercise Testing With Acutely Concussed Adolescent Athletes
Brief Title: Safety Study for Adolescents With Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Barry Willer, Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 030-387696
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Brain Injury; Concussion
MeSH Terms: conditions — Brain Injuries; Brain Concussion | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCTT (Experimental): Participants received an standardized exercise stress test within 7 days of concussive injury. Stress test is stopped when participant experiences any exacerbation of symptoms. Heart rate at time of symptom exacerbation is referred to as the threshold heart rate (THR). Stress test is known as the Buffalo Concussion Treadmill Test.
  Interventions: Other: Exercise stress test (BCTT)
- No BCTT (No Intervention): All participants in the no intervention arm did not get assessed using the BCTT until they had fully recovered or when they had their second clinic visit fourteen days after their first visit.

INTERVENTIONS:
Other: Exercise stress test (BCTT) — Participants are assessed for exercise tolerance using a treadmill with gradually increasing angle to increase workload. Stress test is stopped when there is symptom exacerbation or when participant experiences voluntary exhaustion.
  Arms: BCTT

SUMMARY:
The purpose of the study was to determine if administration of an exercise stress test within the first ten days after a sports related concussion would delay or otherwise interfere with recovery.

DETAILED DESCRIPTION:
The purpose of the study was to determine if administration of an exercise stress test within the first ten days after a sports related concussion would delay or otherwise interfere with recovery. All participants were adolescents injured while playing sports. All concussions were confirmed by an experienced sports medicine physician before random assignment of the participant to receive the treadmill test to determine exercise intolerance or not.

Recovery was defined as (a) return to asymptomatic state; (b) ability to exercise to exhaustion without exacerbation of symptoms and (c) confirmation of recovery by a physician who is blinded to the assignment and to results of exercise testing. Symptoms were self reported on a daily basis using an online data record.

Regardless of recovery rate all participants were assessed at two weeks following their first clinic visit. At the second visit all subjects, regardless of group assignment were assessed on ImPACT, and the treadmill based exercise stress test. Individuals who were not recovered by the second visit were followed until recovered no matter how long that took.

Analysis of data examined recovery rates of the two groups of adolescents to determine whether use of a exercise stress test early after concussion caused any adverse events or interfered in any way with recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with sports related concussion that appear for their first clinic visit within 10 days of injury

Exclusion Criteria:

* Evidence of focal neurologic deficit;
* inability to exercise due to orthopaedic injury;
* diabetes or known heart disease; increased cardiac risk; ADHD; depression; anxiety; history of moderate or severe brain injury; more than 3 prior concussions;
* inability to understand spoken English.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to Full Recovery | 2-168 days
  Asymptomatic; Able to exercise to exhaustion without exacerbation of symptoms, confirmed by examination of a physician blinded to results

CONTACTS AND LOCATIONS:
Overall Officials: John J Leddy, MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willer BS, Haider MN, Bezherano I, Wilber CG, Mannix R, Kozlowski K, Leddy JJ. Comparison of Rest to Aerobic Exercise and Placebo-like Treatment of Acute Sport-Related Concussion in Male and Female Adolescents. Arch Phys Med Rehabil. 2019 Dec;100(12):2267-2275. doi: 10.1016/j.apmr.2019.07.003. Epub 2019 Aug 1. PMID 31377190